CLINICAL TRIAL: NCT00117078
Title: Aranesp® Monthly Preference Study - 2
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Amgen (Industry)
Responsible Party: Global Development Leader, Amgen Inc.
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20020380
Record Dates: First submitted 2005-06-30; First posted 2005-07-04 (Estimated); Last update posted 2008-09-30 (Estimated); Status verified 2008-09

CONDITIONS: Kidney Disease
Keywords: Kidney disease, Renal, CKD (Chronic Kidney Disease); CRI (Chronic Renal Insufficiency), Pre-dialysis, Amgen; Aranesp®, Darbepoetin alfa, QW dosing; Q2W dosing, Q4W dosing; Patient preference, Subject preference
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic; Patient Preference | interventions — Darbepoetin alfa

INTERVENTIONS:
Drug: Aranesp®

SUMMARY:
The purpose of this study was to evaluate subject preference for Aranesp® administered once monthly (i.e., every 4 weeks (Q4W)) or Procrit® administered once weekly (QW).

ELIGIBILITY:
Inclusion Criteria: - Subjects must have signed written informed consent - Be on Procrit® QW or Q2W for a minimum of 8 weeks - Must currently be on a stable dose of Procrit® (defined as less than 25% change in Procrit® dose over the 4 week period immediately prior to enrollment, with no missed doses) - Have Hgb 10-12 g/dL for at least 4 weeks prior to study start - Have 15 less than GFR less than 89 mL/min/1.73 m2 Exclusion Criteria: - Currently receiving investigational erythropoietic agents - Self-injecting at home with Procrit® - Expected to initiate renal replacement therapy (dialysis or transplantation) within 1 year of study start - Have less than 1 year life expectancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

PRIMARY OUTCOMES:
Subject preference

SECONDARY OUTCOMES:
Subject productivity and subject selection of Aranesp® or Procrit® therapy in the parallel arm portion and at study conclusion.

CONTACTS AND LOCATIONS:
Overall Officials: MD, Study Director — Amgen

REFERENCES:
- See also: Notice regarding posted summaries of trial results — http://download.veritasmedicine.com/REGFILES/amgen/Amgen_results_disclaimer.pdf
- See also: To access clinical trial results information click on this link — http://download.veritasmedicine.com/REGFILES/amgen/08D_FDAMA_113_Posting_Summary_33_NESP_20020380.pdf
- See also: FDA-approved Drug Labeling — http://www.aranesp.com/
- See also: AmgenTrials clinical trials website — http://www.amgentrials.com